CLINICAL TRIAL: NCT05720143
Title: Evaluation of Clinical and Radiographic Outcomes of Immediate Dental Implants After Using Three Bone Splitting Techniques in Narrow Mandibular Alveolar Ridges: A Randomized Controlled Clinical Study
Brief Title: Evaluation of Dental Implants After Using Several Bone Splitting Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-OMFS-01-2023
Record Dates: First submitted 2023-01-28; First posted 2023-02-09 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Jaw, Edentulous
Keywords: Osseodensification; Piezosurgery; Magnetic mallet
MeSH Terms: conditions — Jaw, Edentulous | interventions — Piezosurgery

STUDY DESIGN:
Who Masked: Participant
Masking Description: Blinding Participant and Statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Osseodensification group: (Experimental): Ridge splitting and expansion were carried out by creating horizontal and vertical cuts with piezosurgery, followed by expansion of the alveolar ridge using osseodensification burs
  Interventions: Procedure: Osseodensification
- Magnetic mallet group: (Experimental): Ridge splitting and expansion were performed using piezosurgery to create horizontal and vertical cuts, followed by chisels with a magnetic mallet to expand the ridge
  Interventions: Procedure: Magnetic mallet
- Piezo-surgery group (Experimental): Ridge splitting and expansion were performed with piezosurgery inserts, followed by bone expanders
  Interventions: Procedure: Piezo-surgery

INTERVENTIONS:
Procedure: Osseodensification — Procedure: Two horizontal and one vertical osteotomies will be performed using piezosurgery, followed by ridge expansion with osseodensification burs. Immediate implant placement will then be performed.
  Arms: Osseodensification group:
Procedure: Magnetic mallet — Procedure: Two horizontal and one vertical osteotomies will be performed using piezosurgery, followed by ridge expansion using chisels with a magnetic mallet. Immediate implant placement will then be performed.
  Arms: Magnetic mallet group:
Procedure: Piezo-surgery — Two horizontal and one vertical osteotomies will be performed using piezosurgery, followed by ridge expansion using piezosurgery inserts and bone expanders. Immediate implant placement will then be performed.
  Arms: Piezo-surgery group

SUMMARY:
In both complete and partial tooth loss, the use of dental implants as artificial replacements for missing teeth is a well-established and effective treatment modality, leading to high patient satisfaction and improved quality of life (1).

Horizontal deficiencies of the alveolar ridge can hinder implant-supported rehabilitation due to insufficient bone volume to support implant dimensions, negatively affecting the final prosthetic outcome from both functional and esthetic perspectives (2).

The split-crest technique reduces treatment time, the number of required surgical procedures, and the risk of complications, making it more acceptable to patients. Additionally, it allows for dental implant placement during the same surgical procedure and eliminates the need for a donor site for graft harvesting (3).

In this study, patients with posterior tooth loss in a narrow mandibular ridge underwent dental implant rehabilitation following alveolar ridge splitting and expansion performed using osseodensification, piezosurgery, or a magnetic mallet.

DETAILED DESCRIPTION:
The objective of this study is to compare ridge width gain following ridge splitting and expansion with simultaneous implant placement using osseodensification, piezosurgery, or a magnetic mallet in individuals with narrow mandibular alveolar ridges.

Thirty-nine patients will be randomly allocated into three groups. In Group 1, ridge splitting and expansion will be performed using piezosurgery and bone expanders, followed by simultaneous implant placement.

In Group 2, osseodensification burs will be used after ridge splitting, with simultaneous implant placement.

In Group 3, a magnetic mallet will be used after ridge splitting, with simultaneous implant placement.

ELIGIBILITY:
Inclusion Criteria:

1. Patients able to attend follow-up appointments.
2. Alveolar ridges with sufficient height for the placement of a standard dental implant.
3. Presence of spongy bone with at least 1 mm of width between the cortical plates.
4. Absence of systemic or local conditions that could affect bone metabolism.

Exclusion Criteria:

1. Severe concavity on the vestibular or palatal side of the alveolar ridge.
2. Uncontrolled periodontal disease.
3. History of radiotherapy in the head and neck region.
4. Smokers or patients with parafunctional habits.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-06-28 (Actual)

PRIMARY OUTCOMES:
The marginal bone loss | Assessments will be conducted 4 months after surgery and 6 months after functional loading.
  Changes in bone height following ridge splitting and expansion were assessed radiographically. Measurements were performed using cone beam computed tomography (CBCT) and periapical radiography
The bone width gain radiographically | At baseline, after surgery, 4 months after surgery, and 6 months after functional loading.
  The extent of bony expansion represents the increase in alveolar ridge width in the buccolingual direction, as determined by radiographic assessment using CBCT.

SECONDARY OUTCOMES:
Implant stability quotients (ISQ) | Measurements will be taken at the time of surgery and again 4 months postoperatively.
  The Implant Stability Quotient (ISQ), measured using the MEGA device, provides a numerical assessment of both primary and secondary stability of dental implants. The scale ranges from 1 to 100, with higher values indicating greater stability and a higher likelihood of successful osseointegration.
Insertion Torque | During the surgical procedure.
  The implant insertion torque was measured during implant placement using a dental implant torque wrench and recorded in Newton-centimeters (N·cm).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Albassal, MSc, Principal Investigator — Department of Oral and Maxillofacial Surgery, University of Damascus Faculty of Dentistry, Damascus; Munir Harfouch, MSc PhD, Study Director — Department of Oral and Maxillofacial Surgery, University of Damascus Faculty of Dentistry, Damascus; Mazen Zenati, MSc PhD, Study Director — Department of Oral and Maxillofacial Surgery, University of Damascus Faculty of Dentistry, Damascus
Locations (1):
- University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pozzi A, Mura P. Immediate Loading of Conical Connection Implants: Up-to-2-Year Retrospective Clinical and Radiologic Study. Int J Oral Maxillofac Implants. 2016 Jan-Feb;31(1):142-52. doi: 10.11607/jomi.4061. PMID 26800171
- [Background] Chiapasco M, Zaniboni M, Boisco M. Augmentation procedures for the rehabilitation of deficient edentulous ridges with oral implants. Clin Oral Implants Res. 2006 Oct;17 Suppl 2:136-59. doi: 10.1111/j.1600-0501.2006.01357.x. PMID 16968389
- [Background] Bassetti MA, Bassetti RG, Bosshardt DD. The alveolar ridge splitting/expansion technique: a systematic review. Clin Oral Implants Res. 2016 Mar;27(3):310-24. doi: 10.1111/clr.12537. Epub 2015 Jan 14. PMID 25586966
- [Background] Buser D, Mericske-Stern R, Bernard JP, Behneke A, Behneke N, Hirt HP, Belser UC, Lang NP. Long-term evaluation of non-submerged ITI implants. Part 1: 8-year life table analysis of a prospective multi-center study with 2359 implants. Clin Oral Implants Res. 1997 Jun;8(3):161-72. doi: 10.1034/j.1600-0501.1997.080302.x. PMID 9586460
- [Background] Cochran DL, Buser D, ten Bruggenkate CM, Weingart D, Taylor TM, Bernard JP, Peters F, Simpson JP. The use of reduced healing times on ITI implants with a sandblasted and acid-etched (SLA) surface: early results from clinical trials on ITI SLA implants. Clin Oral Implants Res. 2002 Apr;13(2):144-53. doi: 10.1034/j.1600-0501.2002.130204.x. PMID 11952734